CLINICAL TRIAL: NCT05594628
Title: The Effects of Neuromuscular Training on Peroneal Eccentric Strength, Fatigue and Functional Performance in Young Women Basketball Players
Brief Title: Perturbation Based Neuromuscular Training Effects on Peroneal Strength, Fatigue and Functional Performance Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozge Kocaer, Research Assistant/Physiotherapist, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1108799
Record Dates: First submitted 2022-10-11; First posted 2022-10-26 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Healthy Young Women; Basketball Players

STUDY DESIGN:
Intervention Model Description: After first evaluation groups are randomly assigned to 2 groups. Both groups keep attending basketball trainings. One group is just going to keep attending basketball trainings, one group is going to keep attending usual basketball trainings and going to receive neuromuscular training that will be added in warming up exercises
Who Masked: Participant
Masking Description: Adolescent female basketball players that is not currently doing any prevention programme and not currently injured in last 6 months that will make them not to attend any training that happened
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training+Basketball training (Experimental): After all participiants are evaluated, they will be divided randomly to two groups, which one group will be taking neuromuscular training+usual basketball training
  Interventions: Other: Neuromuscular training
- Control group(Basketball training) (No Intervention): After all participiants are evaluated, they will be divided randomly to two groups, which one group will be taking just the usual basketball training and not any extra interventions.

INTERVENTIONS:
Other: Neuromuscular training — Neuromuscular training is designed as 8 weeks and 2 times a week, and approximately 20 minutes per session for Neuromuscular training+usual basketball training group. Other group is only going to keep attending usual basketball training.
  Neuromuscular training consisted 3 exercises:
  First exercise is passing the ball to side to side on bosu with standing on one leg. 60-90 seconds on time, 30-60 seconds off time. 2 sets for both passing sides and bilaterally.
  Second exercise is standing on bosu unilaterally and while standing stabilized, switching basketball hand to hand as dribbling on the floor. Exercise will be on for 60-90 seconds and off for 30-60 seconds, 2 sets for each side Third exercise is jumping with one stance/leg, and landing with double stance while a therabant is attached to the belly and pulling with a minimum/medium force from one side. Changing legs after one jump, 6 times for both side is equal to 1 set of the exercise. It will be done 2 sets for both sides.
  Arms: Neuromuscular Training+Basketball training

SUMMARY:
In the literature neuromuscular exercise programs are often used for prevention in sport players. Literature lacks of perturbation exercises and its effects on peroneal's muscle strength, fatigue and individual's performance parameters. This study will investigate if it is possible to achieve improvements on peroneal eccentric strength, fatigue, dynamic balance and individual's performance with the exercises mainly based on side perturbations.

DETAILED DESCRIPTION:
Chronic ankle instability is very common in adolescent female basketball players. In the literature neuromuscular exercise programs are often used for prevention in sport players that usually contains of strength and/or balance exercises. Perturbation exercises are oftenly used in sport players for returning the sport or prevention but literature lacks of its effects statistically. This study will investigate if it is possible to achieve improvements on peroneal eccentric strength, fatigue, dynamic balance and individual's performance with the exercises mainly based on side perturbations. Strength and fatigue evaluations will be made with Cybex dynanometer. Dynamic balance evaluations will be made with Y-Balance Tests. Individual's performance parameter evaluations will be made with vertical jump test, cross jump test and side hop test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-injured within the 6 months female basketball players that are willing to join the research

Exclusion Criteria:

* That has a injury within 6 months with missing trainings at least 2 times in a row or having vestibuler dysfunction

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Changes in Peroneal eccentric strength | 10 weeks
  Force will be evaluated with Cybex Humac NORM, as Nm/kg(Newton-meters/kg). At 30° /s speed, 3 trials will be made with submaximal force for participants to understand the movement. After trials 4 maximal strength repetition will be made. Highest repetition, and average of 4 repetition will be used for analysis. Before and after the intervention evaluation will be made.
Changes in Peroneal endurance parameters | 10 weeks
  Endurance will be evaluated with Cybex Humac NORM, as Nm/kg(Newton-meters/kg). At 180° /s speed, 5 trials will be made with submaximal force for participants to understand the movement. After trials 20 maximal strength repetition will be made. Endurance is described as containing strength for a duration of time, it can be evaluted with Fatigue index/Endurance parameters will be evaluated with comparing last 10 repetion to first 10 repetion to assess the difference. Before and after the intervention evaluation will be made.

SECONDARY OUTCOMES:
Changes in Dynamic Balance | 10 weeks
  It will be evaluated with Y Balance test to anterior, posteromedial, posterolateral sides. The distance will be recorded with cm's. Before and after the intervention evaluation will be made.
Changes in Cross Hop Test | 10 weeks
  It will be evaluated through cross jumping 3 times on a 6 meter-line. The distance will be recorded wtih cm's. Before and after the intervention evaluation will be made.
Changes in Vertical Jump Test | 10 weeks
  It will be evaluated with Takei Jumpmeter. The height of the jump will be recorded with Takei Jumpmetre with cm's. Before and after the intervention evaluation will be made.
Changes in Side Hop Test | 10 weeks
  2 lines with 30 cm distance will be placed. Players will complete 10 jumping from side to side without stepping on the lines. Unsuccessfull jumps will be excluded. The time will be recorded with chronometer. Before and after the intervention evaluation will be made.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem University, Istanbul
  - Istanbul University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gribble PA, Robinson RH. Alterations in knee kinematics and dynamic stability associated with chronic ankle instability. J Athl Train. 2009 Jul-Aug;44(4):350-5. doi: 10.4085/1062-6050-44.4.350. PMID 19593416
- [Background] Taylor JB, Ford KR, Nguyen AD, Terry LN, Hegedus EJ. Prevention of Lower Extremity Injuries in Basketball: A Systematic Review and Meta-Analysis. Sports Health. 2015 Sep-Oct;7(5):392-8. doi: 10.1177/1941738115593441. Epub 2015 Jun 26. PMID 26502412
- [Background] Mendez-Rebolledo G, Guzman-Munoz E, Gatica-Rojas V, Zbinden-Foncea H. Longer reaction time of the fibularis longus muscle and reduced postural control in basketball players with functional ankle instability: A pilot study. Phys Ther Sport. 2015 Aug;16(3):242-7. doi: 10.1016/j.ptsp.2014.10.008. Epub 2014 Nov 7. PMID 25869423
- [Background] Kim KM, Hart JM, Saliba SA, Hertel J. Modulation of the Fibularis Longus Hoffmann Reflex and Postural Instability Associated With Chronic Ankle Instability. J Athl Train. 2016 Aug;51(8):637-643. doi: 10.4085/1062-6050-51.10.05. Epub 2016 Sep 1. PMID 27583692
- [Background] Asadi A, Saez de Villarreal E, Arazi H. The Effects of Plyometric Type Neuromuscular Training on Postural Control Performance of Male Team Basketball Players. J Strength Cond Res. 2015 Jul;29(7):1870-5. doi: 10.1519/JSC.0000000000000832. PMID 25563677
- [Background] Benis R, Bonato M, La Torre A. Elite Female Basketball Players' Body-Weight Neuromuscular Training and Performance on the Y-Balance Test. J Athl Train. 2016 Sep;51(9):688-695. doi: 10.4085/1062-6050-51.12.03. Epub 2016 Nov 8. PMID 27824252
- [Background] Eils E, Schroter R, Schroder M, Gerss J, Rosenbaum D. Multistation proprioceptive exercise program prevents ankle injuries in basketball. Med Sci Sports Exerc. 2010 Nov;42(11):2098-105. doi: 10.1249/MSS.0b013e3181e03667. PMID 20386339
- [Background] Hurd WJ, Chmielewski TL, Snyder-Mackler L. Perturbation-enhanced neuromuscular training alters muscle activity in female athletes. Knee Surg Sports Traumatol Arthrosc. 2006 Jan;14(1):60-9. doi: 10.1007/s00167-005-0624-y. Epub 2005 Jun 4. PMID 15937713